CLINICAL TRIAL: NCT04274855
Title: Effect of Trait Anxiety in Women on Oral Health Status and Oral Health Care-Seeking Behavior: A Cross-Sectional Study
Brief Title: Effect of Trait Anxiety in Women on Oral Health Status and Oral Health Care-Seeking Behavior
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mariam Ayman Amin Sharaf, Principal investigator, Ain Shams University
Other Study IDs: 830
Record Dates: First submitted 2020-02-16; First posted 2020-02-18 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Anxiety Disorders; Oral Disease; Periodontal Diseases; Periodontal Attachment Loss; Periodontal Pocket; Periodontal Inflammation; Gingival Recession; Gingival Bleeding; Gingival Diseases; Bruxism; Caries,Dental; Health Care Seeking Behavior; Health Care Utilization; Self-Perception
Keywords: Trait anxiety; Oral health; Oral health status; Oral health outcomes; Periodontal; Gingival; Caries risk assessment; Bruxism; Healthcare utilization; Health care-seeking behavior; Perceived oral health
MeSH Terms: conditions — Anxiety Disorders; Mouth Diseases; Periodontal Diseases; Periodontal Attachment Loss; Periodontal Pocket; Gingival Recession; Gingival Hemorrhage; Gingival Diseases; Bruxism; Dental Caries; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Trait anxiety is the tendency of an individual to perceive environmental stimuli such as different events and situations as threatening; it's stable and reflects how an individual generally feels.

In 2015, it was estimated that 3.6% of the population lived with anxiety disorders globally, i.e. approximately 264 million people lived with anxiety disorders worldwide of which 31.36 million resided in the Eastern Mediterranean region, that's to say, 10% of the global number of anxiety cases. Moreover, females were more affected than males in a proportion of 4.6% as opposed to 2.6% respectively. The prevalence of anxiety has increased by 14.9% from 2005 to 2015. In addition, in 2017, approximately 42 million new cases were recorded globally.

In Egypt, the total number of anxiety cases were more than 3 million in 2015 thus indicating that 4.2% of the total population lived with anxiety.

Anxiety may affect the individual's utilization of dental services and predispose to a delay in seeking dental treatment and thus might compromise the overall oral health.

Accordingly, this study aims to investigate the effect of trait anxiety on the oral health status of women and determine their behavior towards the utilization of dental services.

To our knowledge, no previous research has been conducted to assess such relationship in Egypt.

DETAILED DESCRIPTION:
Trait anxiety is a major risk factor for developing anxiety disorders and major depressive disorder, all sharing the same genetic and environmental etiological factors. Another hypothesis is that the etiological factors predispose first to the occurrence of trait anxiety which afterwards, develops into anxiety disorders and clinical depression. Based on this, it's of great importance to be attentive to trait anxiety in clinical practice and research. It's also important to investigate how trait anxiety leads to poorer health outcomes in order to lower its burden and consequences.

Years lived with disability (YLD) is one component that assists in measuring the burden of disease. YLD is the number of years that a person lives with disease. Globally, 24.6 million years lived with disability was due to anxiety disorders. 354 YLD per 100,000 populations were recorded in the Eastern Mediterranean region. Moreover, anxiety ranked the seventh cause of YLD in the Eastern Mediterranean region.

Oral disorders (e.g. periodontal disease and dental caries) collectively have been the most prevalent conditions from 1990 to 2017. Globally, 3.4 billion people lived with oral disorders in 2017.

Bruxism by definition is an activity that involves clenching and grinding of the teeth during sleep(nocturnal bruxism) or when awake(diurnal bruxism). Dentists regard bruxism as a major issue due to its consequences, which range from the destruction of the tooth structure and dental restorations to tempro-mandibular joint (TMJ) manifestations as well as temporal headaches reported by the patients. Psychological disorders such as stress and anxiety are risk factors for the development of bruxism in individuals. Results from previous studies on the relationship between anxiety and bruxism were contradictory; while some studies reported an association between anxiety in different age groups and bruxism, other studies denied such relationship. It's important to study the association between common mental disorders and the occurrence of bruxism activity.

High frequency of sugar consumption in food and beverages has been linked to several common mental disorders. Individuals with mood disorders usually follow a diet that has high amounts of sugar and fats and low amount of fibers. Dental caries is majorly dependent on the frequency of sugar intake, in addition to its form and amount. Therefore individuals with common mental disorders are at an increased risk of developing 'rampant caries'. Rampant caries by definition is a progressive and rapidly appearing dental caries with acute onset, which leads to early pulp involvement, and affects a large number of erupted teeth. Therefore it is of great importance for dental practitioners not only to treat the disease outcome, but also to identify the different phases of the disease. According to this, assessing the risk of developing dental caries in mentally vulnerable patients has been of great importance to tailor a preventive approach specially designed for each patient.

Study procedures:

* A comprehensive literature review was conducted using electronic databases to identify relevant tools (questionnaires and clinical examination tools) to be used in the present study.
* Data about socio-demographic characteristics, severity of trait anxiety(assessed by Egyptian version of State-Trait Anxiety Inventory (STAI Y2 form), presence of bruxism activity, self-perceived dental health status and oral health care-seeking behavior will be collected by means of questionnaires.
* Clinical examination to assess periodontal health condition and caries risk assessment will be conducted.
* All data, as well as, clinical examination will be conducted via one well-trained investigator.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian women
* Age range: From late adolescence to early elderly (20-55 years of age)

Exclusion Criteria:

* Women who do not consent to participate in the study.
* Women who have any diagnosed medical disorders that directly affect their oral health (e.g. Diabetes).
* Women with any diagnosed mental disorders. (Due to the increased incidence of dental caries and gingival disease in addition to the side effects of psychotropic drugs).
* Pregnant women. (Due to the affection of gingival and periodontal condition).
* Women seeking dental treatment.(Otherwise, oral health care-seeking behavior will be biased).

Their number will be reported by a flow chart.

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: A convenient sample of Egyptian women attending Faculty of Dentistry, Ain Shams University for reasons other than seeking dental treatment (e.g. accompanying other patients) will be recruited and enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Estimated)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Presence of gingival and periodontal disease | February 2020-November 2020
  Community Periodontal Index(CPI) on a scale that ranges from 0 to 4, where 0 indicates healthy gingival condition and 4 indicates unhealthy gingival condition (periodontitis)
Risk of developing dental caries | February 2020-November 2020
  American Dental Association (ADA) caries risk assessment tool adult form
Reports of bruxism activity | February 2020-November 2020
  Self-reported questionnaire which includes six questions with good content and face validity to assess bruxism activity on a 4-point Likert scale.
  This questionnaire was translated into Arabic language in the current study. This questionnaire is conducted in the form of an interview.

SECONDARY OUTCOMES:
Oral health care-seeking behavior | February 2020-December 2020
  Five self-reported English questions adopted from previous studies for the same purpose. Those questions were translated into Arabic language in the current study.
  This questionnaire is conducted in the form of an interview.
Self-perceived dental health status | February 2020-December 2020
  Participants are asked to rate their dental health status on 6-point scale from 'excellent' to 'very poor'.

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Sharaf, Masters, Principal Investigator — Ain Shams University; Amira Badran, PhD, Study Director — Ain Shams University; Reham Abou ElFadl, PhD, Study Director — Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Kesim S, Unalan D, Esen C, Ozturk A. The relationship between periodontal disease severity and state-trait anxiety level. J Pak Med Assoc. 2012 Dec;62(12):1304-8. PMID 23866479
- [Background] Kisely S, Sawyer E, Siskind D, Lalloo R. The oral health of people with anxiety and depressive disorders - a systematic review and meta-analysis. J Affect Disord. 2016 Aug;200:119-32. doi: 10.1016/j.jad.2016.04.040. Epub 2016 Apr 21. PMID 27130961
- [Background] Sandi C, Richter-Levin G. From high anxiety trait to depression: a neurocognitive hypothesis. Trends Neurosci. 2009 Jun;32(6):312-20. doi: 10.1016/j.tins.2009.02.004. Epub 2009 May 4. PMID 19409624
- [Background] Winocur E, Uziel N, Lisha T, Goldsmith C, Eli I. Self-reported bruxism - associations with perceived stress, motivation for control, dental anxiety and gagging. J Oral Rehabil. 2011 Jan;38(1):3-11. doi: 10.1111/j.1365-2842.2010.02118.x. PMID 20557433
- [Background] Restrepo CC, Vasquez LM, Alvarez M, Valencia I. Personality traits and temporomandibular disorders in a group of children with bruxing behaviour. J Oral Rehabil. 2008 Aug;35(8):585-93. doi: 10.1111/j.1365-2842.2007.01838.x. Epub 2008 Apr 15. PMID 18422509
- [Background] Parish CL, Feaster DJ, Pereyra MR, Alcaide M, Cohen M, Levin S, Gustafson D, Merenstein D, Aouizerat B, Donohue J, Webster-Cyriaque J, Wingood G, Kempf M, Metsch LR. Dental insurance, dental care utilization, and perceived unmet dental needs in women living with HIV: Results from the Women's Interagency HIV Study. J Public Health Dent. 2019 Dec;79(4):343-351. doi: 10.1111/jphd.12336. Epub 2019 Aug 16. PMID 31418877
- [Background] Ainamo J, Barmes D, Beagrie G, Cutress T, Martin J, Sardo-Infirri J. Development of the World Health Organization (WHO) community periodontal index of treatment needs (CPITN). Int Dent J. 1982 Sep;32(3):281-91. No abstract available. PMID 6958657